CLINICAL TRIAL: NCT06367205
Title: Norepinephrine Infusion Combined With Goal-directed Fluid Therapy Reduces Delayed Graft Function Incidence in Patients Undergoing Kidney Transplantations: a Randomized Multicenter Clinical Trial
Brief Title: Norepinephrine Infusion Combined With Goal-directed Fluid Therapy in Patients Undergoing Kidney Transplantations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LY2023-135-A
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Delayed Graft Function; End Stage Renal Disease; Kidney Transplantation
Keywords: Norepinephrine; Goal-directed fluid therapy; Randomized controlled trial
MeSH Terms: conditions — Delayed Graft Function; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-Directed Fluid Therapy (GDFT) group (Experimental): Following anesthesia induction, patients will be connected to the FlowTrac/Vigileo monitoring system to facilitate the recording of pertinent hemodynamic parameters, including stroke volume variation (SVV), stroke volume, and cardiac output. Then, Norepinephrine Infusion Combined with Goal-directed Fluid Therapy will be administered. Efforts are made to sustain a mean arterial pressure (MAP) of ≥ 80 mmHg.
  Interventions: Drug: Goal-Directed Fluid Therapy (GDFT)
- Regular Fluid Therapy group (Active Comparator): Patients will not undergo monitoring with the FlowTrac/Vigileo system throughout the whole procedure. Anesthesiologists will rely on their clinical expertise and intraoperative circulatory hemodynamic assessment to regulate fluid infusion rates and administer medications as necessary to sustain a mean arterial pressure (MAP) of ≥ 80 mmHg until the conclusion of the surgical procedure.
  Interventions: Drug: Regular Fluid Therapy

INTERVENTIONS:
Drug: Goal-Directed Fluid Therapy (GDFT) — Norepinephrine will be administered intravenously at a rate of 0.06 µg/kg/min, followed by the implementation of fluid therapy guided by SVV until reaching our target. In instances where SVV ≤ 13%, indicative of adequate effective circulating blood volume, the fluid infusion rate will be adjusted to 1 ml/kg/h. Conversely, if SVV > 13%, denoting inadequate effective circulating blood volume, a rapid infusion of 1 ml/kg of crystalloid fluid will be administered over 2 minutes, with subsequent observation of fluid reactivity after a further 2-minute interval. This process is reiterated until SVV ≤ 13% is attained. Should SVV > 13% recurs during surgery, the aforementioned intervention is repeated.
  Other Names: GDFT
  Arms: Goal-Directed Fluid Therapy (GDFT) group
Drug: Regular Fluid Therapy — Anesthesiologists will rely on their clinical expertise and intraoperative circulatory hemodynamic assessment to regulate fluid infusion rates and administer medications as necessary
  Arms: Regular Fluid Therapy group

SUMMARY:
Delayed graft function (DGF), delineated by the necessity for dialytic intervention within the initial week post-transplantation, afflicts approximately 20%-50% of recipients. The primary objective of this study is to investigate the potential efficacy of norepinephrine infusion in conjunction with goal-directed fluid therapy (GDFT) in mitigating the occurrence of DGF among individuals undergoing kidney transplantations. The findings of this investigation have the potential to advance the field of perioperative care in kidney transplantations by providing insights into optimized management strategies.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) presents a formidable challenge to global healthcare systems. With ongoing advancements in surgical techniques, kidney transplantation has emerged as a principal therapeutic modality for individuals afflicted with end stage renal disease (ESRD), markedly enhancing their long-term prognosis and overall quality of life postoperatively. Nevertheless, the occurrence of delayed graft function (DGF) represents a prevalent early complication following kidney transplantations, mainly stemming from the ischemia-reperfusion injury incurred by the transplanted kidneys and the utilization of extended criteria donor organs. The manifestation of DGF can precipitate primary allograft nonfunction, acute rejection episodes, and potentially fatal outcomes. Vigilant attention to perioperative fluid management emerges as a cornerstone in mitigating the risk of DGF. Recent strides in goal-directed fluid therapy (GDFT) have garnered substantial attention within critical care contexts, with empirical evidence underscoring its favorable impact on postoperative outcomes in critically ill cohorts. However, the efficacy of GDFT specifically in the context of kidney transplantation remains a subject of ongoing debate and scrutiny. Hence, the imperative arises to investigate potential strategies aimed at attenuating the incidence of DGF in this patient demographic.

ELIGIBILITY:
Inclusion Criteria:

1. Recipients aged 18 years or older
2. Scheduled to undergo kidney transplantations under general anesthesia
3. Cadaveric kidney transplantations
4. Sign the informed consent form

Exclusion Criteria:

1. Donors aged under 18 years
2. Donor kidneys classified as Maastricht category I or II
3. Contraindications to radial artery catheterization
4. Pregnancy
5. Cardiac dysfunction (exercise tolerance less than 4 METS)
6. Severe liver dysfunction (Child Pugh C-grade)
7. Respiratory diseases with tidal volume intolerance exceeding 8ml/kg
8. Severe arrhythmias, including atrial fibrillation, frequent atrial or ventricular premature beats, moderate or severe aortic and mitral regurgitation
9. Double-kidney transplantations
10. Simultaneous organ or additional surgeries during kidney transplantations
11. Repeat kidney transplantations
12. Concurrent participation in other clinical trials
13. Patients deemed ineligible by researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of delayed graft function (DGF) | Patients will be followed from postoperative day 1 to 7.
  The need for dialytic intervention within the initial week post-transplantation

SECONDARY OUTCOMES:
The area under the curve of serum creatinine levels from postoperative day 1 to 7 | Patients will be followed from postoperative day 1 to 7.
  The area under the curve of serum creatinine levels from postoperative day 1 to 7
Duration of DGF | Patients will be followed from surgery completion to the last dialysis up to 84 days post-surgery.
  The interval from surgery completion to the last dialysis up to 84 days post-surgery
Number of dialysis sessions during postoperative hospitalization | Patients will be followed from surgery completion to discharge，an average of 20 days.
  Number of dialysis sessions during postoperative hospitalization
Total urine output on the second postoperative day | Patients will be followed on the second postoperative day.
  Total urine output on the second postoperative day
Duration of intensive care unit (ICU) stay | Patients will be followed during Intensive care unit (ICU) stay, an average of 2 days.
  Duration of intensive care unit (ICU) stay
Length of hospitalization | Patients will be followed from hospitalization to discharge, an average of 20 days.
  Length of hospitalization
Incidence of readmission within 30 days post-discharge | Patients will be followed from discharge to 30 days after discharge.
  Incidence of readmission within 30 days post-discharge

OTHER OUTCOMES:
The incidence of acute rejection during hospitalization | Patients will be followed from surgery completion to discharge, an average of 20 days.
  The incidence of acute rejection during hospitalization
The survival rates of transplanted kidneys at the one-year postoperative mark | Patients will be followed from surgery completion to one year after surgery.
  The survival rates of transplanted kidneys at the one-year postoperative mark
The survival rates of transplanted patients at the one-year postoperative mark | Patients will be followed from surgery completion to one year after surgery.
  The survival rates of transplanted patients at the one-year postoperative mark
The occurrence of adverse events (AEs) | Patients will be followed from surgery completion to discharge, an average of 20 days.
  The occurrence of adverse events (AEs) recorded by the common terminology criteria for adverse events (CTCAE) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Principal Investigator — Department of Anesthesiology Renji Hospital
Locations (3):
- China (3):
  - the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - General Hospital of Northern Theatre Command, Shenyang, Liaoning
  - Renji Hospital, Shanghai, Shanghai Municipality